

# The Effectiveness of Peer-to-Peer Community Support to Promote Aging in Place

Protocol Number: 000001

**Protocol Version Date**: 4/17/2016

**Coordinating Center**: University of Wisconsin

Study PI: Elizabeth A. Jacobs, MD MAPP

800 University Bay Drive

Suite 210

Madison, WI 53705

Study Coordinator: Rebecca Schwei

Funding Sponsor: Patient Centered Outcomes Research Network (PCORI)

# **Sub-Investigators at Research Sites**

1. Paul Castro: Jewish Family Service

3580 Wilshire Boulevard

Seventh Floor

Los Angeles, CA 90010

(323) 761-8800

2. Kali Deyoung: Community Place of Greater Rochester

145 Parsells Ave. Rochester, NY 14609

(585) 327-8839

3. Jenni Frumer: Alpert Jewish Family and Children's Service

5841 Corporate Way

Suite 200

West Palm Beach, FL 33407

(561) 684-1991

4. Laura Pinsoneault Alliance for Strong Families and Communities

11700 W Lake Park Dr, Milwaukee, WI 53224

414-359-6603

# **Table of Contents**

| Recruitment Strategies | 2 |
|---|---|
| Contacting Potential Participants via the Telephone Prior to Enrollment in the Study | 4 |
| Inclusion and Exclusion Criteria | 5 |
| Matching | 5 |
| Enrolling More than One Person per Household | 6 |
| Enrollment in Study | 6 |
| Updating or Changing Participant Information Once Enrolled | 6 |
| Reminder Letter | 7 |
| Reminder Communication at Baseline Survey | 7 |
| Consent and Baseline Visit | 8 |
| Monthly Postcard Reminder | 8 |
| 3 Month Hospital, Emergency Department, and Urgent Care Data Collection via phone | 8 |
| 6 month survey data collection in-person | 9 |
| Reminder Communication for 6 month Survey | 9 |
| 6 month Survey-Data collection via phone | 10 |
| 9 Month Hospital, Emergency Department, and Urgent Care Data Collection via phone | 11 |
| 12 month Endline | 111 |
| Reminder Communication for 12 month Survey | 12 |
| Medical Records Review | 13 |
| Unexpected Circumstances | 13 |
| Exiting the Study | 13 |
| Missing Data Points for a Participant | 14 |
| Reentry into the Study After Exiting | 14 |
| Payment | 14 |
| Appendix | |

Introductory Letter for Participants (Community Place, AJFCS, JFS of LA)

Failed Contact Recruitment Letter (Community Place)

Reminder Letter (Community Place, AJFCS)

Failed Contact 3, 6, 9, 12 month data collection (Community Place)



# **Recruitment Strategies**

#### Community Place

Community Place currently has 210 people receiving peer to peer support and 408 people on the wait list to receive peer to peer support. These numbers are fluid. All people in both groups have access to all other services that community place offers older adults in their community such as access to the Senior Center, various services we can connect with through our caseworker (Home delivered meals, benefits eligibility, Catholic Family Center-Elder one, Food link, Clothing services, legal consulting services, and Life span (Financial Budgeting, caregivers plan, HEP, High Cap-Health Insurance, Elder abuse prevention, and Rep pay program)).

All the people that are in the correct age range (≥65 years old) and have no known cognitive impairment will be uploaded into the study database in DatStat. People receiving peer to peer support will receive ID Numbers R100E to R499E and people receiving standard community services (on the wait list to receive peer to peer support) will receive ID numbers R500C to R999C. The following variables or a subset of these variables will be uploaded for all participants: ID, First Name, Last Name, Mailing Address, Phone, Age, Date of birth, gender, race, language preference, P2P program type, peer companion name, study group, RA first name, RA last name, RA telephone, RA email, Site PI.

- A. One recruitment strategy will be to contact people off of a pre-specified list of people receiving peer to peer support or on the wait list to receive peer to peer support. These people are already receiving community services from Community Place. We will send out letters to the first 10 people on the list. The letter will give them the option to call us but it will also let them know that we will be calling them within the next two weeks to see if they are interested in participating in the research study. Research staff will select the next person to call and recruit to the study in the recruitment pattern according to the matching strategy that the biostatisticians prepared based on the sociodemographic breakdown of the clientele that are currently receiving peer to peer support. We will send out the *Introductory Letter* to potential participants on the wait list and to potential participants currently receiving peer to peer support. We will send out eligibility letters to people enrolled in peer-to-peer support and on the wait list simultaneously. Every 2-3 weeks we will send letters to 10 new people.
- B. A second recruitment strategy will be by making an announcement about the study at monthly training meetings for both Foster grandparent and senior companion programs. After the announcement is made, the research coordinator will approach potential participants at monthly training meetings and ask them if they are interested in learning more. If interested, we will tell them about the study, screen them for eligibility send them home with a consent form and set up a time to conduct the baseline interview. There is the possibility of enrolling 15-20 people at this meeting. This meeting occurs every month.
- C. A third recruitment strategy will be to hold informational sessions for the purpose of recruiting eligible participants for the study creating our "waitlist". These sessions will be held at community centers around town and in other venues where older adults frequent.



D. Community Place will be partnering with Star Program to recruit additional peers.

Recruitment Goal: As of February 23, 2016 the new recruitment goal at Community Place will be to recruit 226 participants into the study (113 experimental and 113 control)

# Alpert Jewish Family and Children's Service

The Alpert Jewish Family and Children's Service, West Palm Beach currently serves approximately 205 people who receive peer to peer support. There is not currently a waiting list so we will be recruiting people out of the community to serve as the control group. All people in both groups have access to all other services that the Jewish Family and Children's Service offers older adults in the community. People receiving peer to peer support will receive ID Numbers PB100E to PB499E and people receiving standard community services (on the wait list to receive peer to peer support) will receive ID numbers PB500C to PB999C.

A list of participants that are currently receiving peer to peer support will be uploaded into DatStat. However, only first name, age, date of birth, gender and race will be uploaded into the system. The Research Staff will keep a separate list of contact information for these participants on a secure file on her computer. Once a participant agrees to be in the study, then the additional contact information (phone number, address, last name) will be added into DatStat.

- A. One recruitment strategy will be to contact people off of a pre-specified list of people receiving peer to peer support. These people are already receiving services from the Jewish Family and Children's Service. We will send out letters to the first 10 people on the list. The letter will give them the option to call us but it will also let them know that we will be calling them within the next two weeks to see if they are interested in participating in the research study. Research staff will select the next person to call based on the number of people they are trying to recruit in each of the pre-specified categories (ex: white women 65-70). The biostatisticians have created a list of the number of people we should recruit in each demographic bucket based on the demographic breakdown of the people currently receiving peer to peer support. We will then send out the *Introductory Letter* to potential participants from the sessions (on the "wait list") and to potential participants currently receiving peer to peer support. We will send out eligibility letters to people enrolled in peer-to-peer support and to those who are eligible for peer to peer services simultaneously. Every 2-3 weeks we will send letters to 20 new people.
- B. We are also going to hold informational sessions for the purpose of recruiting eligible participants for the study creating our "waitlist". These sessions will be held in three adult gated communities Century Village, Golden Lakes and Banyan Springs and also our sister agencies. We will then send out the *Introductory Letter* to potential participants from the sessions (on the "wait list"). Alternatively, we will collect demographic information from participants at the information sessions and if it is feasible we may even conduct screenings on site.

We will send out eligibility letters to people enrolled in peer-to-peer support and to those who are eligible for peer to peer services simultaneously. Every 2-3 weeks we will send letters to 20 new people.



Recruitment Goal: As of September 3, 2015 the new recruitment goal at Jewish Family Services of Palm Beach will be to recruit 300 participants into the study (150 experimental and 150 control)

#### Jewish Family Service of LA

Jewish Family Service of Los Angeles (JFSLA) currently has 57 people receiving peer to peer support and 35 people on the wait list to receive peer to peer support. They are actively expanding their program. All people in both groups have access to all other services that JFSLA offers older adults in their community such as case management, mental health services, link to community resources, meals, and transportation.

A list of participants receiving peer to peer support will be uploaded into DatStat

- A. One recruitment strategy will be to contact people off of a pre-specified list of people receiving peer to peer support or on the wait list to receive peer to peer support. These people are already receiving community services from JFS of LA. We will send out letters to the first 10 people on the list. The letter will give them the option to call us but it will also let them know that we will be calling them within the next two weeks to see if they are interested in participating in the research study. Research staff will select the next person to call and recruit to the study in the recruitment pattern according to the matching strategy that the biostatisticians prepared based on the sociodemographic breakdown of the clientele that are currently receiving peer to peer support. We will send out the *Introductory Letter* to potential participants on the wait list and to potential participants currently receiving peer to peer support. We will send out eligibility letters to people enrolled in peer-to-peer support and on the wait list simultaneously. Every 2-3 weeks we will send letters to 10 new people.
- B. A second recruitment strategy will be to recruit from Park LaBrea and/or meal programs that are put on by JFS of LA.

<u>Recruitment Goal:</u> As of February 23, 2016 the new recruitment goal at Jewish Family Services of Los Angeles will be to recruit 60 participants into the study (30 experimental and 30 control).

Contacting Potential Participants via the Telephone Prior to Enrollment in the Study (If we are unable to reach a potential participant via telephone, we will leave the following message.)

Hello {U:DATSTAT\_FIRSTNAME}. My name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I am calling to see if you would like to participate in a survey research study to better understand what helps older adults stay in their homes and communities. If you are interested in learning more about the Aging in Place study please call me back at {U:RA\_TELEPHONE} and leave me a message if I'm not at my desk. Otherwise, I will call you back in one week to talk with you. If you are not interested in receiving any more calls from me about this study, please call me and let me know and I will not contact you again. Again, my name is {U:RA\_FIRST} and my phone number is {U:RA\_TELEPHONE} and I look forward to talking with you soon. Have a great day.

We will call back in one week for our second attempt and leave the same message. On the third phone call attempt one week later, we will leave the following message.



Hello {U:DATSTAT\_FIRSTNAME}. My name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling again to see if you would like to participate in the research study about helping older adults stay in their homes and communities. If you are interested in learning more about the Aging in Place study please call me back at {U:RA\_TELEPHONE} and leave me a message if I'm not at my desk. I will not be reaching out to you again about this study. Again, my name is [U:RA\_FIRST] and my phone number is [U:RA\_TELEPHONE] and I hope to talk with you soon. Have a great day.

After the third failed attempt, we will send them the Letter after 3<sup>rd</sup> attempt Failed Recruitment Control or Letter after 3<sup>rd</sup> attempt Failed Recruitment Experimental. All attempts to contact a participant will be documented in DatStat with outcome of the call.

If the research staff talks with a participant but "now is not a good time" then the research staff and the potential participant should set up a better time to talk, whether that is tomorrow or next month. In this situation, the research staff should consider this contact attempt still open (i.e. if this is the first attempt than the first attempt stays open). It is only when you don't reach a participant that the contact attempt closes and we move on to the next contact attempt.

The first time the research staff successfully connects with a participant in person or via the telephone they will follow the screening script outlined in the screening survey.

#### Inclusion & Exclusion Criteria

Inclusion Criteria

- ≥ 65
- Eligible for peer to peer companion services
- Living independently or in independent care

#### Exclusion Criteria

- Receives > 40 hours of in home care from someone other than spouse
- Has plans to move to a higher level of care in the next year
- Has a score on the telephone interview of cognitive status (TICS) ≤ 25
- Doesn't live permanently in one location "snow birds"

If in the peer to peer group the following exclusion criteria also apply

- Utilization of a peer companion is temporary
- Primary reason older adult has a peer companion is to provide respite for their caregiver

#### Matching

For Community Place and Alpert Jewish Family and Children's Service (AJFCS), we are matching participants on the following characteristics: age group (<70, 70-80, and ≥ 80 years), gender (male and female), race/ethnicity (African American, Hispanic, and non-Hispanic White) and at Community Place we are also matching based on County (Monroe or Livingston).

At both all sites we are going to recruit people from the waiting list and match them with people already receiving peer to peer services. Every month research staff at UW will ask to see the matching spreadsheet as a way to monitor how matching is progressing at each site.

#### Enrolling more than one person per household (added 1/14/2016)

As of February 22, 2016, we will only enroll one person per household. This is the protocol for determining which person from the household we will enroll.

- a. If Participant A is enrolled in the study (signed the consent form) and they say they would like their partner would like to participate, the research staff person will let them know that according to study protocol we are only allowed to enroll one person per household. Participant A will be the person that is enrolled in the study.
- b. If prior to enrollment a study staff person is informed that both partners in a couple want to participate in the study. The staff person will let the two participants know that we can only enroll one participant from the couple. If we only need one person then the research staff will screen and enroll that person.
- c. If we know in advance there is a couple interested in participating and both people are needed for the study then we will randomly select one person per household. In this case you should screen both participants. If both participants are deemed eligible to participate you should first assign one participant heads and one participant tails. Then you should pull out the randomization envelope and open it. This envelope will tell you which participant you will enroll. At this time you will discard the envelope.

#### **Enrollment in Study**

Enrolling people in the study is a three step process. Step 1, is technically a pre-screen, we only want to upload people into DatStat who we think are eligible. If for whatever reason we find out that they are not eligible then we don't want them in the database. You can email Becky and she will delete their entry from DatStat. It is also a good idea for all RAs to keep a list of participants that have been deleted to ensure that you don't accidentally contact them again. Step 2 is the formal screening. If during the formal screening it turns out that they are not eligible then DatStat marks them as ineligible, and they will be removed from your workflow. They do not need to be formally exited from the study. Step 3 is when they sign the consent form during the baseline survey. Once they sign the consent form then, they are officially enrolled in the study. Moving forward, if for whatever reason the person withdraws consent, dies or meets a main study outcome that would be when you officially exit them from the study using the exit survey. The rule of thumb is we only exit people from the study who are officially enrolled, and people are only officially enrolled once they sign the consent form.

# Updating or changing participant information once enrolled in study

When updating or changing participant information in Discovery, you can update participant information however you like, including assigning someone to the most accurate study group, prior to the participant signing the consent form. Once a participant signs a consent form, at that time we will consider all the information entered in Discovery to be updated and accurate. At this point some very critical variables such as study arm, race, age, gender, site, language, DOB, can never be changed, even if they are wrong. If at any time after the participant signs a



consent, you realize there is an error in one of these data categories you cannot change the information in Discovery but rather you need you to record that information in a participant log (a word document that you will keep on your computer) and you need to alert Becky of the change. Every few months Becky will ask for a copy of these participant logs. The participant log should include the Participant ID number, the person who made the change in the DatStat system, the original incorrect value and the new corrected value.

If at some point you realize that you made an error in updating information, you need to let Becky know and she will consult with the UW research team to figure out how to move forward.

# Reminder Letter (if participant indicates they would like one)

After baseline visit is scheduled reminder letter with copy of the consent form is sent to participant. It is up to the research staff to determine if they would like to just send the reminder letter or if they would like to send the reminder letter with the consent form.

#### **Reminder Communication for Baseline Survey**

Research staff can place the reminder call whenever they think makes the most sense. Some people prefer to place a reminder call the day before and then also call the participant in the morning to confirm that they are still planning on the appointment. Other staff may prefer to call the participant the morning of the appointment. Regardless of timing, there needs to be at least one reminder phone call placed and logged in DatStat. Research staff can feel free to log all of their contact calls but at a minimum they need to log one contact.

#### Phone call if talking to a person

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to remind you that I have an appointment set up with you to do your baseline survey for the Aging in Place Study. The appointment is at {U:BASELINE\_LOCATION} on {BASELINE\_DATE}. Does this time still work for you?"

If yes, "Is there anything special I need to know about getting access to where you live? Will I need to go through a security gate, or use a buzzer to let you know I have arrive?" (make note of anything the relevant the participant says) "Great, I look forward to seeing you soon. Please call me if you have any questions. My phone number {U:RA\_TELEPHONE} and my name is {U:RA\_FIRST} {U:RA\_LAST}"

A. If no, ask them if we can find another time to set up the appointment. Research staff works to set up a time for the baseline survey. Change in appointment date is documented in DatStat.

#### Phone call-voicemail

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE} and I was calling to remind you that I have an appointment set up with you to do your baseline survey at {U:BASELINE\_LOCATION} at {U:BASELINE:DATE} for the Aging in Place Study. If this time still works for you I do not need a call back. If you have decided you would no longer like to



participate in the study or would like to change your appointment time please feel free to give me a call back. My phone number is {U:RA\_TELEPHONE}. Thanks and have a nice day. "

#### **Consent and Baseline Visit**

Please refer to the baseline survey documents for instructions on completing the baseline visit. Once participants sign the consent form they are officially enrolled in the study and this is considered time zero for that participant.

# **Monthly Postcard Reminders**

We will send generic thank you and reminder postcards on the first of the month to all participants who are active in the study at months 2, 5, 8, 11. The postcard will thank them for being in the study and will remind the participant to please mark down the times they go the hospital, emergency department and urgent care on their calendars. The postcard will also include the contact information for the study staff.

Thank you for continuing to participate in the Aging in Place Study. Don't forget to mark down all the times you stay overnight in the hospital, visit the emergency room or go to urgent care on your study calendar. We look forward to talking with you very soon. (Card will have study staff phone number)

**3 Month Hospital, Emergency Department, and Urgent Care Data Collection via phone** The window to complete the three month data collection on time is 2 weeks before the 3 month anniversary and 2 weeks after the 3 month anniversary. The window will close 6 weeks after the 3 month anniversary.

If we are unable to reach a potential participant, we will leave a message.

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from{U:DATSTAT:SITE}. I was calling to talk to you about the Aging in Place study. I would like to ask you a few questions for your 3 month survey so please give me a call back. If you have decided you would no longer like to participate in the study please call me with that information as well. Again this {U:RA\_FIRST} {U:RA\_LAST} from{U:DATSTAT:SITE}. and my phone number is{RA\_TELEPHONE}. Thanks and have a nice day. "

We will call back in one week for our second attempt and leave the same message. We will call back in one week for our third attempt and leave the same message but it will be our last attempt to reach that participant via phone. If no success after the third attempt DatStat will trigger a letter. The letter is titled *Letter after 3<sup>rd</sup> attempt to contact for data collection*. All attempts to contact a participant will be documented in DatStat with outcome of the calls documented as well.

For questions and procedures related to 3 month data collection, please refer to the 3 month telephone survey document.

6 month survey data collection in-person



A participant is eligible to complete the sixth month survey 2 weeks before and 2 weeks after but data collection will be allowed 8 weeks after the 6 month anniversary.

# Scheduling 6 month Survey

Call participant 1 month before sixth month anniversary and say the following.

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to set up a time to meet with you in person so we can do our next survey for the Aging in Place study." Set up a time to meet with the participant in person and document in DatStat.

If we are unable to reach a potential participant, we will leave a message.

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to set up a time to meet with you in person so we can do our next survey for the Aging in Place study. If you could call me back so I can schedule a time for us to meet, my number is {U:RA\_TELEPHONE}. If you have decided you would no longer like to participate in the study please call me with that information as well. Again this is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. and my phone number is {U:RA\_TELEPHONE}. Thanks and have a nice day. "

We will call back in one week for our second attempt and leave the same message. We will call back in one week for our third attempt and leave the same message but it will be our last attempt to reach that participant via phone. If no success after the third attempt DatStat will trigger a letter. The letter is titled *Letter after 3<sup>rd</sup> attempt to contact for data collection*. All attempts to contact a participant will be documented in DatStat with outcome of the calls documented as well.

After an appointment is set up the staff will send a reminder letter to participants that request it, confirming the date and time of the appointment. Reminder Letter Document

#### Reminder Communication for 6 month Survey

Research staff can place the reminder call whenever they think makes the most sense. Some people prefer to place a reminder call the day before and then also call the participant in the morning to confirm that they are still planning on the appointment. Other staff may prefer to call the participant the morning of the appointment. Regardless of timing, there needs to be at least one reminder phone call placed and logged in DatStat. Research staff can feel free to log all of their contact calls but at a minimum they need to log one contact.

#### Phone call talking to a real person

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to remind you that I have an appointment set up with you to do our next survey for the Aging in Place study at {U:6MONTH\_LOCATION} at {U:6MONTH\_TIME}. Does this time still work for you?" (Response: Yes, No)



If yes, "Great, I look forward to seeing you soon. Please call me if you have any questions. My phone number is {U:RA\_TELEPHONE} and my name {U:RA\_FIRST} {U:RA\_LAST}.

If no, ask them if we can find another time to set up the appointment. Research staff works to set up a time for the interview. Change in appointment date is documented in DatStat.

#### Phone call- voicemail

"Hi, my name {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to remind you that I have an appointment set up with you to do your sixth month followup survey at {U:6MONTH\_LOCATION} at {U:6MONHT\_TIME} for the Aging in Place Study. If this time still works for you I do not need a call back. If you have decided you would no longer like to participate in the study or would like to change your appointment time please feel free to give me a call back. My phone number is {U:RA\_TELEPHONE}. Thanks and have a nice day. "

# 6 month Survey-Data collection via phone

A participant is eligible to complete the sixth month survey 2 weeks before and 2 weeks after but data collection will be allowed 8 weeks after the 6 month anniversary.

"Hi, my name is U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to see if now would be a good time to ask you a few questions for the sixth month follow up for the Aging in Place Study. Is now a good time to talk?

Yes- ask all questions

No-set up a better time to talk and schedule it in DatStat

If we are unable to reach a potential participant, we will leave a message.

"Hi, my name is U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}.. I was calling to set up a time to talk with you. If you could call me back so I can ask you some questions for the Aging in Place Study, my number is {U:RA\_TELEPHONE}. If you have decided you would no longer like to participate in the study please call me with that information as well. Again this is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE} and my phone number is {U:RA\_TELEPHONE}. Thanks and have a nice day. "

We will call back in one week for our second attempt and leave the same message. We will call back in one week for our third attempt and leave the same message but it will be our last attempt to reach that participant via phone. If no success after the third attempt DatStat will trigger a letter. The letter is titled *Letter after 3rd attempt to contact for data collection*. All attempts to contact a participant will be documented in DatStat with outcome of the calls documented as well.

Please refer to the 6 month survey for instructions on how to complete the 6 month data collection.



**9 Month Hospital, Emergency Department, and Urgent Care Data Collection via phone** Window to complete the nine month data collection on time is 2 weeks before the 9 month anniversary and 2 weeks after the 9 month anniversary. The window will close 6 weeks after the 9 month anniversary.

If we are unable to reach a potential participant, we will leave a message.

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to, as promised the last time we spoke, to ask you information for the Aging in Place study. If you could call me back so I can ask you a few questions I would really appreciate it. My number is {U:RA\_TELEPHONE}. If you have decided you would no longer like to participate in the study please call me with that information as well. Again this is {U:RA\_FIRST} from {U:DATSTAT:SITE} and my telephone number is {U:RA\_TELEPHONE}. Thanks and have a nice day. "

We will call back in one week for our second attempt and leave the same message. We will call back in one week for our third attempt and leave the same message but it will be our last attempt to reach that participant via phone. If no success after the third attempt DatStat will trigger a letter. The letter is titled *Letter after 3<sup>rd</sup> attempt to contact for data collection*. All attempts to contact a participant will be documented in DatStat with outcome of the calls documented as well.

Hello {U:DATSTAT\_FIRST}, This is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. It has been 3 months since I last talked to you as a part of the Aging in Place study. Do you have a minute for me to ask you a few questions? (Yes, No)

- If no, schedule a better time to call back

Please refer to the 9 month survey for instructions on 9 month data collection.

#### 12 month Endline

A participant is eligible to complete the sixth month survey 2 weeks before and 2 weeks after but data collection will be allowed 8 weeks after the 12 month anniversary.

Scheduling 12 month Survey

Call participant 1 month before 12 month anniversary and say the following.

"Hi, my name is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to set up a time to meet with you in person for the final survey of the Aging in Place Study."

Set up a time to meet with the participant in person and document in DatStat.

If we are unable to reach a potential participant, we will leave a message.



"Hi, my name {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to set up a time to meet with you in person for the Aging in Place Study. If you could call me back so I can schedule a time for us to meet, my number is {U:RA\_TELEPHONE}. If you have decided you would no longer like to participate in the study please call me with that information as well. Again this is {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. and my phone number is {U:RA\_TELEPHONE}. Thanks and have a nice day. "

We will call back in one week for our second attempt and leave the same message. We will call back in one week for our third attempt and leave the same message but it will be our last attempt to reach that participant via phone. If no success after the third attempt DatStat will trigger a lette. The letter is titled *Letter after 3<sup>rd</sup> attempt to contact for data collection*. All attempts to contact a participant will be documented in DatStat with outcome of the calls documented as well.

After an appointment is set up the staff will send *Reminder Letter* to participants that request it, confirming the date and time of the appointment.

#### Reminder Communication for 12 month Survey

Research staff can place the reminder call whenever they think makes the most sense. Some people prefer to place a reminder call the day before and then also call the participant in the morning to confirm that they are still planning on the appointment. Other staff may prefer to call the participant the morning of the appointment. Regardless of timing, there needs to be at least one reminder phone call placed and logged in DatStat. Research staff can feel free to log all of their contact calls but at a minimum they need to log one contact.

# Phone call talking to a real person

"Hi, my name {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}. I was calling to remind you that I have an appointment set up with you to do your final 12 month survey for the Aging in Place Study. Your appointment is scheduled for {U:12MONTH\_DATE} at {U:12MONTH\_LOCATION}. Does this time still work for you?"

If yes, "Great, I look forward to seeing you soon. Please call me if you have any questions. My phone number is {U:RA\_TELEPHONE} and my name is {U:RA\_FIRST} {U:RA\_LAST}

If no, ask them if we can find another time to set up the appointment. Research staff works to set up a time for the interview. Change in appointment date is documented in DatStat.

#### Phone call voicemail

"Hi, my name is *name {U:RA\_FIRST} {U:RA\_LAST} from {U:DATSTAT\_SITE}.* I was calling to remind you that I have an appointment set up with you to do your 12 month follow-up survey for the Aging in Place Study. Your appointment is scheduled for {U:12MONTH\_DATE} at {U:12MONTH\_LOCATION}. If this time still works for you I do not need a call back. If you have

Page 12 of 24 Last Updated: 4/17/2016

decided you would no longer like to participate in the study or would like to change your appointment time please feel free to give me a call back. My phone number is {U:RA TELEPHONE}. Thanks and have a nice day. "

Please refer to 12 month survey for instructions on 12 month data collection.

#### **Medical Chart Review**

The purpose of the Medical Chart Review Component of the Study is to see if the number of times participants report visiting the Emergency Department or staying overnight in the Hospital is consistent with what is found in the medical record.

#### Before the next in person visit

Prior to the next in person visit research staff should confirm that the participant signed the consent form for the medical chart review component of the study. If the participant has signed the consent form researcher staff should complete an authorization for release of medical records for the participant. Research staff need to complete the <u>Patient Information section</u> of the form and the <u>date range</u> on the Medical Records to be disclosed section. Research staff should bring two copies of the authorization for release of medical information form to the visit. Research staff should also have a copy of the medical records review form for reference.

# At the in person visit

During the in person visit, at some point the research staff should remind participants about the second component of the study that involves requesting their medical records to confirm that they visited the emergency room and stayed overnight in the hospital on the days that they said they did. Research staff will review the authorization of release of medical information form with the participant and will confirm that the only medical information we are requesting is related to the dates you visited the Emergency Department and the nights the participant spent in the hospital. Research staff will ask participants to sign the authorization of release of medical information form and will leave an extra copy with the participant.

After a participant has signed the Authorization of Release of Medical Information Form Once a participant has signed the release form and once they have completed the study (completed the endline survey or met a main outcome), research staff will copy the authorization file and will keep the original in a locked filing cabinet. They will fax a copy of the authorization form and a cover page (see supporting documents) to the medical records department at every hospital where the participant reported visiting in the last year. We will track the progress of the submission of the requests via our data collection program, DatStat.

#### Follow up with Medical Offices

We will follow up with the medical records department every four weeks to ensure they are processing our request.



#### Receipt of Medical Records

All medical records will be faxed to Dr. Elizabeth Jacobs in Madison, WI. Once we receive a patient's medical record we will enter the dates of hospitalizations and emergency department visits into DatStat using the Medical Record Review Form 1 and Medical Record Review Form 2. All medical records will be kept in a locked drawer in a locked office suite.

#### Accessing medical records for people who have died

If a participant dies prior to us accessing their medical records, we will request the legal guardian or spouse to sign a new form giving us permission to access their medical records.

# Accessing medical records for people who withdraw from the study

If prior to the end of the study a participant withdraws from the study, we will ask them if it is still okay for us to access their medical records. We will remind them that they previously gave us permission to do so and that this will require no additional work on their part. If a participant agrees to this then we will follow the protocol above for accessing medical records.

# **Unexpected Circumstances**

Some trouble shooting situations:

- If the client wants to give you food or drinks politely refuse and stress the quicker we can get the questionnaire done he/she can get back to their regular schedule.
- Participant gets tired in the middle of the questionnaire or you can tell they have lost their attention span to answer the questions. Try to complete study but if not you could try to finish questions over the phone making it easier so you don't have to go back to their homes. Payment will be sent to participant upon completion of the survey if applicable
- If there are interruptions (family comes home, friend comes by to visit, package gets dropped off, etc.) while questionnaire is being asked allow time for the participant to focus back to the task at hand.
- Canceling last minute may be an issue just be sure to make follow up phone calls to reschedule.
- Not home/forgot here the phone call the day before the scheduled time is important so they don't forget you are supposed to come over.
- For the control group a problem we may face is the fact that they don't know who the organization is and we could have higher refusals for that group.

#### **Exiting the Study**

At any time a participant has the right to exit the study. In this case you will answer the following questions on behalf of the participant and then they will not be contacted again for the purposes of the study.

Why is the participant leaving the study? (DATSTAT EXITREASON)

Completed

Deceased

Censored (moved to a higher level of care- i.e. independent care to assisted living)
Unable to Continue (you should mark this answer if the person is too sick to continue)
Unable to Locate



Unwilling to Continue
Withdrawn by study staff
Unknown

What day did this person exit the study? (DATSTAT\_EXITDATE)

What other information should we know about why this person left the study? (DATSTAT EXITCOMMENT)

# Missing Data Points for a Participant

If study staff are not able to contact a participant within the appropriate window of data collection they have not exited the study but this is considered missing data. We will continue trying to contact the participant at every data collection point unless they contact us directly and ask to withdraw from the study. If research staff "miss" a data collection point, they should still try to collect the data but will have to follow the following protocol to ensure data is collected accurately:

Our DatStat workflow set up in your configuration is such that the time point gets updated when EITHER of the following occurs: 1) the survey for that timepoint gets submitted, OR 2) the time point goes out of window. For this participant, the 3 month call went out of window, and thus the timepoint got updated to 6 months.

In order to enter data for the 3 month survey at this point, the following must occur:

- 1. The participant must be edited and their time point set back to "3 months"
- 2. The current open survey (study task = "3 month survey") must be closed by clicking Edit Survey next to the task in the Study Task grid, and changing the status to Final Incomplete
- 3. A new 3 month survey study task must be added. To do this, while in the study Task grid go to the Take Action menu and select Add Survey. Select the survey called "3 month Survey (Ad hoc)". Schedule the survey, and select the Survey Pending status code, and click save. You may now use this task to enter your 3 month data. DO NOT do this until you've done steps 1 and 2.

Any time you make a change like this you need to mark down in your study log that you are making this change and mark down in your survey that this was collected out of window and the reason why. You also need to alert Becky that this change is made and she will record it in the data log,

#### Reentry into the study after exited\*\*

If a participant has exited the study prematurely and contacts study staff about re-entry, the participant is only eligible to participate if

a. They are still within the 1 year follow up period. In this case study staff will begin contacting participant at appropriate time points and other data will be considered missing.

Page 15 of 24 Last Updated: 4/17/2016

- b. They sign a new consent form
- c. PI and Site PI agree to allow him/her to re-enter.

# **Payment**

Completion of baseline= \$25 Completion of sixth month survey = \$25 Completion of endline survey at 12 months = \$50.

# Regular Payment Schedule

Time Zero: \$25 12 Months: \$75

If a participant drops out after 6 months each organization will send the participant the \$25 they have earned.



<sup>\*\*</sup>Participants will never be allowed to collect more than \$100 for participation in the study

# **Appendix**

#### INTRODUCTORY LETTER FOR PARTICIPANTS

#### **Community Place**

October 26, 2015

[Recipient Name]

Dear [Recipient Name]:

My name is Kali DeYoung and I am the Research Assistant for the Aging Services program. I am writing to you today about a great opportunity for you to be a part of a research project we are conducting through the University of Wisconsin.

The purpose of the research is to see if aging in place help older adults live independently in their homes. The information you provide and the results we conclude, will help many people in the future who are in your same situation.

I will be contacting you in the next two weeks (coming weeks) to discuss your participation, conduct a screening and if eligible, set up a time to conduct a baseline interview for this study. You shall receive a small compensation as a token of appreciation for participating in this research project.

I appreciate your consideration and will be happy to answer any questions you may have. I would be grateful if you would call me when you receive this letter even to inform me you are not interested. I can be reached at 585-288-0021 ext. 243 or by email <a href="mailto:kdeyoung@communityplace.org">kdeyoung@communityplace.org</a>. Thank you for choosing [Company Name]. And I look forward to speaking with you about this project.

Sincerely,

Kali DeYoung



#### **AJFCS**

#### Dear Barry

My name is Jenny Madlof and I am the Research Specialist for the Aging Services program at the Alpert Jewish Family and Children's Service in West Palm Beach. I am writing to you today about a great opportunity for you to be part of a research project we are conducting with the University of Wisconsin.

The purpose of the research is to evaluate if aging support programs have the potential to help older adults like you live more independently in your own home. The information you provide and the results we conclude, will help many people in the future who are in the same situation.

I shall be contacting you soon to discuss your participation, conduct a screening and, if eligible, set up a time to conduct a baseline interview for this study. You shall receive a small compensation as a token of appreciation for participating in this research project.

I appreciate your consideration and will be happy to answer any questions you may have. I can be reached at 561-238-0410 or by email at <a href="mailto:jmadlof@jfcsonline.com">jmadlof@jfcsonline.com</a>.

Thank you and I look forward to speaking with you about this project.

Sincerely

Jenny Madlof Research Specialist Peer-to- Peer Aging in Place Study



#### JFS of LA

[Date]

#### Dear [Recipient Name]:

My name is Erika Zambrano-Morales and I am the Research Coordinator for the Senior Health and Wellness Program, an aging services program. I am writing to you today about a great opportunity for you to be a part of a research project Jewish Family Service of Los Angeles is conducting with the University of Wisconsin.

The purpose of the research is to see if social services programs help older adults live independently in their homes. The information you provide and the results we conclude, may help many people in the future who are in your same situation.

I will be contacting you in the coming weeks to discuss your participation, conduct a screening and if eligible, set up a time to conduct an interview for this study. You will receive small financial compensation as a token of appreciation for participating in this research project.

I appreciate your consideration and will be happy to answer any questions you may have. Please feel free to give me a call if you are not interested in participating in this research project or if you have any questions. I can be reached at 213.260.7919 or by email <a href="mailto:ezambrano-morales@jfsla.org">ezambrano-morales@jfsla.org</a>. Thank you and I look forward to speaking with you soon about this project.

Sincerely,

, MA Research Coordinator Senior Health and Wellness Program Jewish Family Service of Los Angeles 3580 Wilshire Blvd Suite 700

Los Angeles, CA 90010 Phone: 213.260.7919 Fax: 323.761.8801

Ezambrano-morales@jfsla.org

www.jfsla.org

tshajirat@jfsla.org www.jfsla.org

Fax: 323.876.6140

7377 Santa Monica Blvd.

West Hollywood, CA 90046

Phone: 323.851.8202 ext. 115

Terry Shajirat, BSW CONNECT Program Coordinator West Hollywood Comprehensive Service Center- Jewish Family Service of Los Angeles

#### **FAILED CONTACT FOR RECRUITMENT LETTER**

# **Community Place**

[Your Name] [Date]

[Recipient Name] [Street Address] [City, ST Zip Code]

# Dear [Recipient Name]:

My name is Kali DeYoung and I am the Research Assistant for the Aging Services program at the Community Place of Greater Rochester. I am writing to you today because I have been unable to reach you by phone to discuss the research project we are enrolling clients into.

Please call or send me an e-mail at your earliest convenience so I can update your information even if you do not want to be a part of the research project. I would be grateful for your call and will be happy to answer any questions or concerns you may have. I can be reached at 585-288-0021 ext. 243 or by email <a href="mailto:kdeyoung@communityplace.org">kdeyoung@communityplace.org</a>. Thank you and I hope to hear from you soon.

Sincerely,

[Your Name] Research Assistant



Last Updated: 11/30/2015

#### **REMINDER LETTERS**

# **Community Place**

[Your Name] 145 Parsells Avenue Rochester, NY 14609 [Date]

[Recipient Name] [Address] [City, ST ZIP Code]

Dear [Recipient Name]:

I am Kali DeYoung, the Research Assistant for the "Aging in Place" study. I am writing to you today to confirm our appointment.

I have an appointment on my calendar for **DATE at TIME**. If this time still works I will see you then but if it isn't a good time please let me know so we can make a new appointment. I can be reached at 585-288-0021 ext. 243 or by email <a href="kdeyoung@communityplace.org">kdeyoung@communityplace.org</a>. (I have also included copies of the consent forms we will discuss and sign during our appointment.)

{**Depends on the person**} Please let me know if you have any questions or concerns. I look forward to meeting with you.

Sincerely,

[Your Name] Research Assistant



# **AJFCS**

Dear Loretta

My name is Jenny Madlof and I am the Research Specialist for the Older Adults Service.of the Alpert Jewish Family and Children's Service in West Palm Beach.. I am writing to you today to confirm our appointment to do the baseline survey for the Aging in Place Research Study.

As agreed upon today, we have an appointment for Monday, October 12, 2015 at 10:00 am in your home. If this time is not suitable, please let me know. I can be reached at 561-238-0410 or by email <a href="mailto:imadlof@jfcsonline.com">imadlof@jfcsonline.com</a>.

I look forward to seeing you soon.

Sincerely,

[Your Name] Research Specialist

# FAILED DATA COLLECTION AT 3, 6, 9 OR 12 MONTHS

# **Community Place**

[Your Name] 145 Parsells Avenue Rochester, NY 14609 [Date]

[Recipient Name] [Street Address] [City, ST ZIP Code]

Dear [Recipient Name]:

Thank you for your participation in the study with [Company Name]. I am writing to you today because I have been unable to reach you by phone or e-mail to complete the next step of our research project. I would be happy to update your information to try and keep everything on track.

Please call or send me an e-mail at your earliest convenience. I would be grateful for your call and will be happy to answer any questions or concerns you may have. I can be reached at 585-288-0021 ext. 243 or by email <a href="mailto:kdeyoung@communityplace.org">kdeyoung@communityplace.org</a>. I look forward to hearing from you.

Sincerely,

[Your Name] Research Assistant

